CLINICAL TRIAL: NCT06583486
Title: A Multi-center, Open-label Study on the Efficacy and Safety of Repeated Treatments With Recombinant Botulinum Toxin Type A for Injection in the Treatment of Moderate to Severe Glabellar Lines
Brief Title: A Study on the Efficacy and Safety of Repeated Treatments With Recombinant Botulinum Toxin Type A for Injection in the Treatment of Moderate to Severe Glabellar Lines
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chongqing Claruvis Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY001-001-Ⅲ-RENEW; CTR20240641 (Registry Identifier: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2024-07-07; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Moderate to Severe Glabellar Lines
Keywords: YY001; Recombinant Botulinum Toxin Type A; Botulinum Toxin; Glabellar Lines
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: Single-arm and long-term follow-up
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Five sites will be repeatedly injected with Rcombinant botulinum neurotoxin type A for injection (YY001) at 0.05 mL each, 2 sites in corrugator muscle of each side and 1 site in the procerus muscle, for a total dose of 20U.The study period is up to 64 weeks, divided into 5 treatment cycles.
  Interventions: Biological: Rcombinant botulinum neurotoxin type A for injection (YY001)

INTERVENTIONS:
Biological: Rcombinant botulinum neurotoxin type A for injection (YY001) — Five sites will be injected at 0.05 mL each, 2 sites in corrugator muscle of each side and 1 site in the procerus muscle, for a total dose of 20U.

SUMMARY:
This is a Multi-center, Open-label Study on the Efficacy and Safety of Multiple Treatments with Recombinant Botulinum Toxin Type A for Injection in the Treatment of Moderate to Severe Glabellar Lines. The study has been designed to evaluate the long-term safety, tolerability, efficacy , maintain time and immunogenicity of multiple treatments with Recombinant Botulinum Toxin Type A for Injection (YY001) in the treatment of moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 65 years (inclusive) at the time of signing the informed consent form.
2. At screening or baseline, participants who complete all visits of the REFINE study without major protocol deviations and SAEs
3. Agree to participate in the study and sign the informed consent form.
4. At the discretion of the investigator, the participants can comply with the protocol requirements.
5. Females and/or males of childbearing potential and their partners: those who should be using effective contraception and have no plans for childbearing, egg donation (females), or sperm donation (males) from the signing of the informed consent form to 3 months after the last administration. female participants of childbearing potential must have had a negative blood pregnancy test (human chorionic gonadotropin) within 7 days prior to the first administration of study drug or a Urine pregnancy test examination must be negative 3 days prior to the first administration of study drug.

Note:

1. Women of childbearing potential are those who have experienced menarche, have not undergone sterilization (hysterectomy or bilateral salpingo-oophorectomy or bilateral tubal ligation), and are not in a state of post-menopausal (defined as absence of menstrual bleeding for 12 months prior to screening, without any other medical reason).
2. Effective contraceptives include: vasectomy, abstinence, intrauterine devices, hormones [oral, patch, ring, injections, implants], barrier methods [diaphragm, cervical cap, sponge, condom].

Exclusion Criteria:

1. Use of medications or treatments prohibited by the REFINE study protocol.
2. Any condition that required permanent discontinuation of study treatment during the REFINE study.
3. Use of nonsteroidal anti-inflammatory drugs including aspirin or anticoagulants within 1 week prior to baseline.
4. Abnormal laboratory tests that, in the assessment of the investigator, are not appropriate for participation in this study: including, but not limited to: alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≥ 2.5 times the upper limit of the normal range (×ULN), creatinine ≥ 2 ×ULN, urea/urea nitrogen ≥ 2 ×ULN.
5. Female who is pregnant or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events and drug-related adverse events during the study. | Up to 64 weeks

SECONDARY OUTCOMES:
The proportion of participants who achieve a score of 0 or 1 on the investigator's assessment of GL severity. | At Weeks 1, 4, 12, 24 (if applicable), and 36 (if applicable) after each treatment.
  Glabellar lines at maximal frown are based on the 4 grade Facial Wrinkle Scale: 0 (none), 1 (mild), 2 (moderate) and 3 (severe).
The proportion of participants who achieve a score of 0 or 1 on the participant's self-assessment and Independent Review Committee's assessment of GL severity photos at maximal frown taken on-site. | At Weeks 1(for participants), 4, 12, 24 (if applicable), and 36 (if applicable) after each treatment.
The respond rate on the investigator's assessment of GL severity at maximal frown. | At Weeks 1, 4, 12, 24 (if applicable), and 36 (if applicable) after each treatment.
  The respond rate: The proportion of participants achieving a score of 0 or 1 and at least a two-grade improvement from the baseline, on the investigator's assessment and the participant's self-assessment concurrently of GL severity at maximal frown.
The proportion of participants with a decrease of at least 1 grade from the baseline, on the investigator's assessment and the participant's self-assessment individually of GL severity at rest. | At Weeks 1, 4, 12, 24 (if applicable), and 36 (if applicable) after each treatment.
  The severity of glabellar lines at rest will be assessed according to the 4 grade scale: 0 (none), 1 (mild), 2 (moderate) and 3 (severe).
Incidence of anti-drug antibodies and neutralizing antibodies during the study. | Up to 64 weeks
The lasting time from a single injection to the participants' score of GL severity at maximal frown on the investigator's assessment return to the baseline. | Up to 64 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wu, Principal Investigator — Peking University First Hospital
Locations (16):
- China (16):
  - Guangdong Second People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xian, Shanxi
  - West China School of Medicine/West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hangzhou First People's Hospital, Westlake University, School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking Union Medical College Hospital , Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Plastic Surgery Hospital, Chinese Academy of Medical Science, Beijing
  - The First Affiliated Hospital of Chongqing Medical University, Hongqing
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No